CLINICAL TRIAL: NCT01241630
Title: Somato-sensory Reflex Arch in Spinal Cord Injury - Effect on Clinical Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-20090113 - 2
Record Dates: First submitted 2010-11-08; First posted 2010-11-16 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2012-10

CONDITIONS: Spinal Cord Injury
Keywords: Somato-sensory reflex arch; Spinal cord injury; Xiao Procedure
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Somatosensory reflex arch (Xiao Procedure) — Cross over surgery. Proximal part of L5 Ventral root is anastomosed to distal part of ventral root of S2 or S3 producing a somato-sensory reflex arch
  Other Names: Somato-sensory reflex arch; Artificial somato-sensory reflex arch

SUMMARY:
Spinal cord injury (SCI) usually affects young people and causes severe bowel and bladder dysfunction. Recently, the concept of a surgically created somat-sensory reflex arch for bladder dysfunction in SCI has been introduced. The concept is promising, not just for bladder but also for bowel dysfunction. However, well designed studies need to be performed before recommending the procedure to a large number of patients worldwide. In this study we perform multidisciplinary studies providing necessary information about the clinical outcome of the somato-sensory reflex arch in adult SCI patients.

The hypothesis is as follows:

1. In a "western setting" the somato-sensory reflex arch can be created in adult SCI patients with only minor morbidity and complications.
2. Somato-sensory reflex arch reduces bladder and bowel symptoms in SCI patients.

DETAILED DESCRIPTION:
Introduction:

Spinal cord injury has a profound impact on the lives of those affected. Quality of life is restricted not only by immobility but also by severe neurogenic bladder and bowel dysfunction. For example, 66% of SCI patients have to empty their rectum digitally, 75% suffer from faecal incontinence and 9% spend more than 60 minutes each time they defecate. Neurological impairment due to SCI is permanent and the average age at injury is only 28 years. The longevity of individuals with SCI is approaching that of the general population and, accordingly, most patients have to live for several decades with severe bladder and bowel symptoms. It is estimated that the number of individuals with SCI in Denmark is 3.000 and each year 10.000 persons in the European Union sustain a SCI. Even though clean intermittent catheterization has successfully reduced mortality due to urinary tract infections or reflux and though several new treatment modalities for neurogenic bowel dysfunction have been introduced, both bladder and bowel dysfunction still rank among the top three causes of impairment of quality of life after SCI.

Somato-sensory reflex arch:

The concept was pioneered by professor Xiao. Animal studies and basic clinical research were performed in the United States and later human clinical studies have been done in Wuhan, China. The surgical procedure principle can briefly be summarized as follows:

All spinal nerves have an anterior efferent root and a posterior afferent root. For the somato-sensory reflex arch (or "Xiao procedure") the posterior (afferent or sensory) root of the 5th lumbar nerve (L5) is kept while the anterior root is cut and anastomosed to the anterior root of a lower segment, usually the third sacral segment (S3). Thereby, a new reflex arch has been created from the skin of the leg through the sensory part of L5 to the spinal cord and further through the anastomosis via S2 or S3 to the bladder and bowel. Strong stimuli at the L5 dermatome, i.e. scratching or electrical stimulation, will then initiate voiding (6,7). Effects of the somato-sensory reflex arch on neurogenic bowel dysfunction have not been studied, but clinical experience indicates that bowel management is substantially facilitated.

The Xiao procedure introduces a completely new concept for management of spinal cord lesions and it has been greeted with optimism worldwide. The number of patients operated in China alone is now more than 3.000 and centres in the United States, Germany and Israel have introduced or modified it. Furthermore, centres in Australia, Finland and Denmark plan to introduce it within the present year. There are, however, serious concerns that need to be addressed:

Clinical follow-up has only been done in very few patients and physiological studies after the procedure are equally few and small.

In spite of the very large number of patients operated in China logistic or cultural factors have prohibited effective follow-up.

A minor improvement in bladder and bowel function may be important to a Chinese patient without access to other treatment but it is unknown whether the Xiao procedure will be an advantage to patients in a western healthcare system.

The mode of action of the somato-sensory reflex arch is very incompletely studied and the mode of action on bowel function not studied at all.

Before the widespread use of somato-sensory reflex arch we find it of utmost importance that well designed studies with validated or even objective endpoints are performed. Results of such studies will have an international impact in either defining indications for a completely new treatment principle or, otherwise, in preventing the widespread use of an ineffective treatment.

Hypotheses:

In March 2009 the core members of our multidisciplinary study team went on a study tour to Wuhan, China. In Wuhan a staggering number of 600 patients had the somato-sensory reflex arch procedure performed in 2008. Based on experience from our visit we pose the following hypotheses:

1. In a "western setting" the somato-sensory reflex arch can be created in adult SCI patients with only minor morbidity and complications.
2. Somato-sensory reflex arch reduces bladder and bowel symptoms in SCI patients.

Patients and Methods:

Spinal cord injured patients

Internationally, two indications for the somato-sensory reflex arch are emerging:

Adult patients with bladder dysfunction due supraconal SCI (above the conus medullaris) and Children with bladder dysfunction due to spinal bifida. Most children with spinal bifida have motor incomplete lesions and, accordingly, the surgical procedure carries a risk of long-lasting or even permanent loss of motor function - typically loss of dorsiflexion of the foot. Whether results from the procedure justify that risk remains to be determined. In contrast, patients with motor complete supraconal SCI, and thereby complete loss of voluntary muscle function below the level of injury, do not run that risk. Therefore, it has been decided that patients in group a) above will be offered the procedure at the Department of Neurosurgery NK, AUH. Initially, 20 patients will undergo the procedure. As the method is new, surgery and follow-up will be performed under strict monitoring with emphasis on neurophysiologic testing and potential complications. Approval will be obtained from the Ethics Committee, patients will be very carefully informed by the neurosurgeon (Dorte Clemmensen) and informed consent will be signed.

Surgical procedure:

The relatively minor surgical procedure has been described in previously. In summary: A hemilaminectomy of L5-S1 is performed. By means of neurophysiology testing the 5th lumbar root and 2nd or 3rd sacral roots are identified on one side. The perineurium is opened and the motor roots are separated from the sensory. The motor roots are transsected and a microanastomosis is created between L5 and S2 or S3. After surgery sprouting occurs and after 12-18 months the reflex arch is functional. Time till clinical effect is therefore also 12-18 months. The advantage of the procedure is that it is performed through a hemilaminectomy of only two segments and the surgical stress in relatively small. The patients are expected to be in their habitual condition within 48 hours.

Post surgical monitoring:

Through informal contacts it has been agreed that complications and basic functional results from three centres about to adopt the procedure (Melbourne, Australia; Helsinki, Finland; and Aarhus, Denmark) will be recorded in a standardized way. Preliminary principles for assessment have been agreed upon and other centres introducing the procedure in the future will be invited to participate. This will allow comparison of results between centres.

Study A). Detailed assessment of functional results of the somato-sensory reflex arch To patients the main concern is whether the procedure is safe and reduces symptoms. Detailed and internationally accepted evaluation forms for adult SCI patients have recently been developed. The so called International Spinal Cord Injury Data Sets have been endorsed by the International Spinal Cord Organisation (ISCoS) and the American Spinal Cord Association (ASIA). Information within the data sets are mainly symptom based but for lower urinary tract function urodynamic assessment is included and for bowel function radiographically determined colorectal transit time is included. From the bowel function data sets the most commonly used scores for bowel dysfunction, including the Neurogenic Bowel Dysfunction Score, developed at our unit, can be computed.

Patients undergoing the surgical procedure will be assessed using the basic and extended lower urinary tract data sets and the bowel function data sets before surgery and 18 months after. Before

Based on the investigations above, we aim at publishing the following sub-studies:

A1). Prospective study of urodynamic function and bladder symptoms before and after somato-autonomic reflex arch in spinal cord injury patients.

A2). Prospective study of colorectal symptoms before and after somato-autonomic reflex arch in spinal cord injury patients.

A3). Prospective study of colorectal transit times and rectal wall properties after somato-autonomic reflex arch in spinal cord injury patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or above with motoric complete
* Spinal cord injury medullary level C4-L4
* Preserved Hamstring reflex (L5)
* Participation acceptance in verbal and writing

Exclusion Criteria:

* Respiratory dependent patient Baclofen pump Malignancy in the urinary tract, surgery on the urinary tract, urethral strictures Ileostomy, Colostomy or radiation towards the area Pregnancy, for men planning a pregnancy with their partner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Urodynamic function and bladder symptoms before and after somato-autonomic reflex arch in spinal cord injury patients | 2013 (anticipated)
  Prospective study of urodynamic function and bladder symptoms before and after somato-autonomic reflex arch in spinal cord injury patients.

SECONDARY OUTCOMES:
Colorectal symptoms before and after somato-autonomic reflex arch in spinal cord injury patients | 2013 (anticipated)
  Prospective study of colorectal symptoms before and after somato-autonomic reflex arch in spinal cord injury patients.
Colorectal transit times and rectal wall properties after somato-autonomic reflex arch in spinal cord injury patient | 2013 (anticipated)
  Prospective study of colorectal transit times and rectal wall properties after somato-autonomic reflex arch in spinal cord injury patients.
Effect of quality of Life after somato-autonomic reflex arch in spinal cord injury patient | 2013 (anticipated)
  Effect of quality of Life after somato-autonomic reflex arch in spinal cord injury patient

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Krogh, MD,PhD, DmSc, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark